CLINICAL TRIAL: NCT03884764
Title: for Patients With Chronic Pelvic Pain Due to Chronic Prostatitis, do Combined Ganglion Impar Denervation and Pulsed Radiofrequency on Sacral Root 3 Acheive Better Analgesia Than Ganglion Impar Alone
Brief Title: Ganglion Impar Denervation and Radiofrequency on Sacral Root 3 for Chronic Prostatic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Diab Fuad Hetta, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SECI-IRB-IORG0009563-724
Record Dates: First submitted 2019-03-20; First posted 2019-03-21 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF on S3 + ganglion impar denervation (Experimental): patients will receive pulsed radiofrequency on sacral root number 3 in conjunction with ganglion impar denervation by alcohol
  Interventions: Procedure: pulsed radiofrequency
- ganglion impar denervation (Active Comparator): patients will receive ganglion impar denervation by alcohol
  Interventions: Procedure: ganglion impar denervation

INTERVENTIONS:
Procedure: pulsed radiofrequency — patients with chronic pelvic pain due to chronic prostatitis will receive pulsed radiofrequency on sacral root number 3 and ganglion impar denervation and the patients will be followed for 6 months to assess pain severity radiofrequency procedure: patients will positioned prone on the operating table and under x-ray guidence sacral foramen number 3 will be identified and through it radiofrequency needle will be advanced to target the sacral root ganglion impar procedure: under x-ray guidance the sacrococcygeal junction is identified and spinal needle will be introduced through it to target ganglion impar and 4 ml of alcohol 50% will be injected
  Arms: PRF on S3 + ganglion impar denervation
Procedure: ganglion impar denervation — patients with chronic pelvic pain due to chronic prostatitis will receive ganglion impar denervationand and the patients will be followed for 6 months to assess pain severity ganglion impar procedure: under x-ray guidance the sacrococcygeal junction is identified and spinal needle will be introduced through it to target ganglion impar and 4 ml of alcohol 50% will be injected
  Arms: ganglion impar denervation

SUMMARY:
the authors will evaluate the added analgesic benefit of pulsed radiofrequency on sacral root 3 with ganglion impar denervation on chronic pelvic pain due to chronic prostatitis

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic pelvic pain due to chronic prostatitis for at least 3 months
* VAS pain score more than 5
* failed analgesic drug treatment

Exclusion Criteria:

* coagulopathy
* neurogenic bladder
* infection at site of procedure

Ages: 16 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
the percentage of patients that achieve more than 50% change of their initial pain on VAS pain score | patients will be evaluated at 3 months postoperatively
  VAS pain is a scale of pain measurements scored grom 0 to 10 in which 0 = no pain and 10 the worst pain immaginable

CONTACTS AND LOCATIONS:
Locations (1):
- Diab, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No